CLINICAL TRIAL: NCT02142972
Title: Low Back Pain Disability, Intensity and Widespread Pain and Relationship to Postpartum Depression
Brief Title: Low Back Pain and Depression: Cohort Study
Status: Completed | Type: Observational
Sponsor: Universidad Rey Juan Carlos (Other)
Responsible Party: Principal Investigator, Josue Fernandez Carnero, PhD, Associate Professor, Universidad Rey Juan Carlos
Other Study IDs: 2011/28
Record Dates: First submitted 2014-05-07; First posted 2014-05-20 (Estimated); Last update posted 2014-05-20 (Estimated); Status verified 2014-05

CONDITIONS: Low Back Pain; Pelvic Pain; Depression
Keywords: Low back pain; Oswestry questionnaire; Post-partum Depression; Pelvic pain
MeSH Terms: conditions — Low Back Pain; Pelvic Pain; Depression; Depression, Postpartum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aims of this study are to investigate whether pelvic pain and low back pain disability are associated with postpartum depression and to compare the prevalence between women without Low back pain and disability and women with Low Back Pain (LBP) and disability every trimester, and correlate postpartum Depression and some clinical and biopsychosocial variables: subgroups of LBP, disability, pain intensity, pain widespread and nationality, in a cohort of Spanish women at 2 months postpartum.

DETAILED DESCRIPTION:
295 pregnant women will formed the cohort, during all pregnancy and two months after delivery. The Edinburgh Postnatal Depression Scale was used to evaluate depressive symptoms at 2 months postpartum. The LBP will be evaluated based on self-administrated questionnaire, and the patients with LBP will be classified in to lumbopelvic groups according to mechanical assessment of the lumbar spine, pelvic pain provocation tests, standard history, pain intensity on visual analogue scale, spread of pain through pain drawings and Oswestry index was used to evaluated the disability. Logistics regression analysis will performed to explain the predictors of depression.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria were being pregnant between for 12 weeks to 16 weeks,
* With an expected normal pregnancy (as determined by midwife),
* Being able to understand and read Spanish.

Exclusion Criteria:

* Exclusion criteria were end of pregnancy before gestational weeks 37 (delivery or abortion),
* Serious intellectual impairment,
* Having had a systemic disease (spondylitis, infectious, vascular, metabolic or endocrine related process), rheumatic disease, fibromyalgia, lumbopelvic pain or
* Verified diagnosis of spinal problems in the previous 6 months, or
* A history of fracture, neoplasm or previous spinal, pelvic or femur surgery.
* Another exclusion criterion was a diagnosis of depression or anxiety in the previous year.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The cohort comprised all pregnant women who were registered consecutively at this primary health care center
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2011-10; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Post-Partum Depression | change from baseline in postpartum depression at 2 months after delivery
  Depressive Symptoms is assessed through the Edinburgh Postnatal Depression Scale (EPDS) (translation - Spanish). It´s a 10-item self-report scale specifically designed to screen for postpartum depression. The scale rates the intensity of depressive symptoms present within the previous 7 days. A cutoff score of ≥10 in the tests is to be used for screening purposes in primary care. When selecting this threshold the sensitivity for detection of major depression increased to almost 100% and the specificity to 82%. The participants filled it in at the first visit and two months postpartum.

SECONDARY OUTCOMES:
Pain Scores in the visual analogue scale | Participants will be followed for the duration of pregnant up to 36 weeks
  The Visual Analog Scale (VAS) is used to assess pain intensity (0-100 mm, where "0" corresponded to "no pain" and "10" to the worst imaginable pain).All participants were evaluated during all their pregnancy: in the first trimester (for 12 to 16 weeks), in the second trimester (for 22 weeks) and in the third trimester (for 36 weeks)
Low back pain disability | Participants will be followed for the duration of pregnant up to 36 weeks
  Disability is measured with the Oswestry Low Back Pain and Disability Questionnaire (ODQ) to compare the prevalence between women without LBP and disability and women with LBP pain and disability every trimester. All participants were evaluated of low back disability during all their pregnancy: in the first trimester (for 12 to 16 weeks), in the second trimester (for 22 weeks) and in the third trimester (for 36 weeks).
Pain drawing area | Participants will be followed for the duration of pregnant up to 36 weeks
  Participants completed detailed pain drawings representing a human body (American Academy in Physical Medicine and Rehabilitation. 2001) to assess pain location (lumbar, pelvic and symphysis pubis). To score the spread of pain, these human body views are uniformly divided into a total of 220 squares, each measuring 0.5 x 0.5 cm. .

CONTACTS AND LOCATIONS:
Overall Officials: Josue Fernandez-Carnero, PhD, Principal Investigator — Universidad Rey Juan Carlos